CLINICAL TRIAL: NCT03113669
Title: An Investigation of Appetitive Cognitive Control: Impact on Treat Outcomes for Binge Eating
Brief Title: Project BITE: Binge Intervention Target Effectiveness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1608004727
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Binge-Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (CBT-GSH) (Other): Participants will receive a clinical intake (1 hour) and 6-sessions (approximately 25 minutes each) over 12 weeks of individual guided self-help CBT for eating disorders based on the treatment approach developed by Dr. Christopher Fairburn to use his self-help book Overcoming Binge Eating with the therapeutic guidance of clinician. Participants will be provided with a copy of Overcoming Binge Eating. The treatment is a largely behavioral treatment that focuses on helping patients engage in more regular eating, reduce dieting behaviors, and eliminate behaviors that contribute to binge eating. All participants in the study will receive the same treatment.
  Interventions: Behavioral: CBT-GSH

INTERVENTIONS:
Behavioral: CBT-GSH

SUMMARY:
The primary aim of this study is to determine how inhibitory neurobiological and neurocognitive processes relate to binge eating treatment outcome.

DETAILED DESCRIPTION:
Binge eating disorder (BED) is characterized by reoccurring binge eating episodes that consist of eating a subjectively or objectively large amount of food over a period of time accompanied by a sense of loss control over eating, in the absence of recurrent compensatory behaviors (e.g., purging). Cognitive behavioral therapy (CBT) is the current gold-standard treatment for reducing binge eating episodes in BED patients. The first-line of recommended CBT treatment is a self-guided intervention called CBT-Guided Self-Help (CBT-GSH). However, for a substantial minority of patients, CBT-GSH fails to reduce binge episodes after treatment. Preliminary findings of the literature suggests that individuals with BED possess deficits in inhibitory control as it relates to food-stimuli. We are studying how inhibitory neurobiological and neurocognitive processes relate to binge eating treatment outcome.

This study involves a brief phone screen and research assessment (approximately 5 hours) to determine eligibility. Eligible participants will receive CBT-GSH, which will include a one-hour clinical intake followed by 6 therapy sessions (approximately 30 minutes each). Participants will also complete research assessments at mid-treatment, post-treatment, and 3 month follow-up intervals. Research assessments include a battery of questionnaires, computerized tasks, interviews, and a task using functional Near Infrared Spectroscopy (fNIR) imaging.

ELIGIBILITY:
Inclusion Criteria:

* Speak, write, and understand English
* Body Mass Index (BMI) of 30 kg/m2 or greater
* Experience objectively or subjectively large binge eating episodes once per week or more for the past three months
* If applicable, have stable psychiatric medication for the past three months
* For the optional ecological momentary assessment, participants must own a smartphone compatible with PACO mobile application

Exclusion Criteria:

* Currently engage (in past three months) in any regular compensatory behaviors (e.g., self-induced vomiting, laxative/diuretic use)
* Acute suicide risk
* Are currently receiving psychological treatment for binge eating
* Are currently receiving weight loss treatment
* Co-morbid clinically significant psychological disorder that would require attention beyond the study treatment (e.g., psychotic disorder, substance dependence)
* Diagnosis of intellectual disability or autism spectrum disorder
* History of neurological condition or traumatic brain injury
* Current pregnancy
* History of bariatric surgery
* Are currently using a stimulant medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Eating Disorder Examination (EDE) | Change from baseline to 3-month follow-up
  The Eating Disorder Examination is a widely utilized, semi-structured interview for the assessment of eating disorder symptoms and the binge-eating module will be used to determine binge episode frequency.

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parker MN, Burton Murray H, Piers AD, Muratore A, Lowe MR, Manasse SM, Ayaz H, Juarascio AS. Prefrontal cortex activation by binge-eating status in individuals with obesity while attempting to reappraise responses to food using functional near infrared spectroscopy. Eat Weight Disord. 2023 Mar 30;28(1):34. doi: 10.1007/s40519-023-01558-z. PMID 36995567